CLINICAL TRIAL: NCT03466489
Title: Prevention of Surgical Site Infections in Total Joint Arthroplasty: Iodine Impregnated Adhesive Drapes Versus Cyanoacrylate-Based Sealant
Brief Title: Floraseal Versus Iodine Impregnated Adhesive Drapes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant were enrolled
Sponsor: University of Miami (Other)
Collaborators: Osteoremedies (Industry)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Assistant Professor, Arthroplasty & Joint Reconstruction, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180222
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Surgical Site Infection; Surgical Wound Infection
Keywords: total joint arthroplasty
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Floraseal (Experimental): The surgical site will first be cleaned with isopropyl alcohol. Once the site is dry, alcohol based chlorhexidine gluconate preparatory solution will be applied to the surgical site. Once dry, the FloraSeal surgical preparatory solution will be applied per the manufacturers recommendations. The extremity will be draped in sterile fashion however adhesive drapes over the surgical site itself will not be applied.
  Interventions: Device: Floraseal
- Control (No Intervention): The operative site is first cleaned with isopropyl alcohol. Once the site is dry, alcohol based chlorhexidine gluconate preparatory solution will be applied to the surgical site. The operative site will then be draped in sterile fashion. An iodine impregnated adhesive drape will then be applied to the surgical site.

INTERVENTIONS:
Device: Floraseal — FloraSeal is a cyanoacrylate-based sealant used in the prevention of surgical site infections.
  Arms: Floraseal

SUMMARY:
Infection after total joint arthroplasty can have devastating consequences. Adhesive drapes have been traditionally used at our institution to help reduce the risk of wound contamination and infection by superficial skin flora. Our primary objective is to determine if a cyanoacrylate-based sealant (FloraSeal microbial sealant) is superior to conventional iodine impregnated drapes in prevention of both superficial and deep surgical site infections in total joint arthroplasty (TJA) patients. A prospective, randomized controlled model will be used to answer this question.

DETAILED DESCRIPTION:
Demand for Total Knee Arthroplasty (TKA) and Total Hip Arthroplasty (THA) is increasing steadily and is projected to continue trending upwards in the coming years. Postoperative infections are a common but also potentially devastating complication of total joint arthroplasty.

Various strategies are employed both pre-operatively and post-operatively to prevent this complication. A 2011 Cochrane Review concluded that Iodine impregnated adhesive drapes had no impact on surgical site infection rate when used in various surgical procedures not specific to orthopaedics. The recent SSI prevention guidelines by the World Health Organization did not find any evidence to support the use of adhesive drapes during surgery and recommends against its use.

Currently, iodine impregnated adhesive drapes in conjunction with either chorahexadine gluconate or Iodine Povacrylex and Isopropyl Alcohol are the standard of care at our institution.

FloraSeal is a cyanoacrylate-based sealant. A cyanoacrylate microbial sealant minimizes endogenous bacteria spread to the surgical site by forming a sterile film bonded onto a patient's skin. This film, which is formed upon polymerization, prevents the spread of microorganisms. The protective mechanism is mechanical: the film traps and immobilizes microorganisms that survive on a patient's skin. It has been previously shown to effectively immobilize both gram positive and gram negative bacteria. Additionally, the sealant itself can effectively reduce the superficial bacterial burden on the skin surface and also helps reduce skin moisture buildup on skin.

Furthermore, with conventional adhesive drapes, the edges must be peeled back at the time of skin closure in order to effectively close the surgical site. It is at this moment that the incision becomes most vulnerable to penetration by local microorganisms. FloraSeal and other cyanoacrylate based sealants remain on the skin for 5 to 10 days until the superficial skin sloughs off.

Studies on sterile pig skin demonstrated FloraSeal to be more effective alone at immobilizing bacteria than incisional drapes. The efficacy was the same when FloraSeal was used with or without the incisional drapes, demonstrating that it may be used as a substitute.

Additionally, a 2013 retrospective study in revision shoulder arthroplasty demonstrated a potential reduction in positive intraoperative deep tissue cultures when using a cyanoacrylate-based microbial sealant versus the iodine impregnated incisional drapes. The study lacked sufficient power to reach significance, calling for further investigation of this effect.

Cyanoacrylate has been investigated in other surgical interventions. A 2008 prospective, randomized multicenter clinical trial in patients undergoing elective open hernia repair demonstrated cyanoacrylate-based microbial sealant independently reduced wound contamination over the course of the operation.

Due to the potentially devastating complications associated with postoperative infection, the investigators seek to find alternative methods of prevention of surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Have signed the written informed consent form

Exclusion Criteria:

* Patients not fluent in the language of the informed consent form
* Prisoners
* Pregnancy
* Reported to have mental illness or belonging to a vulnerable population
* History of dermatitis or allergic reaction to cyanoacrylate based materials or iodine
* Patients undergoing revision total joint arthroplasty secondary to infection
* Allergy to Iodine.
* Patients undergoing total joint arthroplasty in the setting of acute trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Appearance of Surgical Site | 90 days from date of surgery
  The surgical incision will be checked post-operatively for signs of infection or dehiscence.

SECONDARY OUTCOMES:
Intra-operative cultures | Intra-operative - Cannot be clearly defined as it will depend on the duration of the surgical procedure.
  Five wound cultures will be obtained at various points during the operation to test for contamination of the surgical site
Post-operative complication - Antibiotic administration | 90 days from date of surgery
  Some surgical site infections may be managed with either intravenous or oral antibiotics. Both groups will be followed to see if either required antibiotic administration.
Post-operative complication - Re-operation | 90 days from date of surgery
  Some surgical site infections require surgical debridement. Patients will be followed to determine which patients require re-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The researchers will share aggregate data but no individual's data will be shared. De-identified graphs of the accelerometer or range of motion output recordings from the devices may be used to illustrate the device's application.

REFERENCES:
- [Background] Prince D, Kohan K, Solanki Z, Mastej J, Prince D, Varughese R, et al. Immobilization and death of bacteria by Flora Seal® microbial sealant. International Journal of Pharmaceutical Science Invention. 2017 Jun;6(6):45-9.
- [Background] Zhang S, Ruiz R. FloraSeal® microbial sealant: a comprehensive solution to skin flora. 2015.
- [Background] Lorenzetti AJ, Wongworawat MD, Jobe CM, Phipatanakul WP. Cyanoacrylate microbial sealant may reduce the prevalence of positive cultures in revision shoulder arthroplasty. Clin Orthop Relat Res. 2013 Oct;471(10):3225-9. doi: 10.1007/s11999-013-2854-5. PMID 23471553
- [Background] Towfigh S, Cheadle WG, Lowry SF, Malangoni MA, Wilson SE. Significant reduction in incidence of wound contamination by skin flora through use of microbial sealant. Arch Surg. 2008 Sep;143(9):885-91; discussion 891. doi: 10.1001/archsurg.143.9.885. PMID 18794427
- [Background] Bailey IS, Karran SE, Toyn K, Brough P, Ranaboldo C, Karran SJ. Community surveillance of complications after hernia surgery. BMJ. 1992 Feb 22;304(6825):469-71. doi: 10.1136/bmj.304.6825.469. PMID 1547415
- [Background] Webster J, Alghamdi A. Use of plastic adhesive drapes during surgery for preventing surgical site infection. Cochrane Database Syst Rev. 2015 Apr 22;2015(4):CD006353. doi: 10.1002/14651858.CD006353.pub4. PMID 25901509
- [Background] Fairclough JA, Johnson D, Mackie I. The prevention of wound contamination by skin organisms by the pre-operative application of an iodophor impregnated plastic adhesive drape. J Int Med Res. 1986;14(2):105-9. doi: 10.1177/030006058601400210. PMID 3699240
- See also: Product information sheet — https://osteoremedies.com/wp-content/uploads/2017/08/FloraSeal-Sales-Sheet.pdf